CLINICAL TRIAL: NCT02539121
Title: Influence of Acupuncture in the Postpartum Blood Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Principe de Asturias (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RenMai6
Record Dates: First submitted 2015-08-26; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Postpartum Women
Keywords: Labor; Acupuncture; Postpartum hemorrhage; Placental expulsion time; Postpartum blood loss
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): In the intervention group with real acupuncture, after the umbilical cord is clamped, the acupuncturist disinfects the abdominal area with antiseptic and pricks the needle in the point Ren Mai 6. This point is located on the anterior midline, between the umbilicus and the upper part of the pubic symphysis, at a distance of 0.3d from the umbilicus, being d the distance from the umbilicus to the upper part of the pubic symphysis. A sterilized steel needle of 0.25x40 mm is inserted in this point at 15-30 mm, depending on the adipose tissue of the woman. After that, the needle is covered with a opaque plastic cup and the cup is fixed with the adhesive tape.
  Interventions: Device: Acupuncture
- Control (Placebo Comparator): In the control group the puncture of the Ren Mai 6 is not performed, the acupuncturist disinfects the abdominal area with antiseptic and put the needle in the area of Ren Mai 6 without puncturing, after that, the needle is fixed but not punctured, and it is covered with a opaque plastic cup fixed with adhesive tape, guaranteeing that neither the mother nor the midwife responsible of measuring the variables can identify the assigned group.

INTERVENTIONS:
Device: Acupuncture — Acupuncture needles
  Arms: Acupuncture

SUMMARY:
In this study, a single blind randomized trial with third party evaluation is carried out in order to compare the postpartum blood loss when Ren Mai 6 point is stimulated and when this point is not stimulated.

Investigators focus on measuring the volume of postpartum blood during the third stage of labor and during the first two hours after birth. A significant reduction in the volume of bleeding would imply a reduction in the rate of postpartum hemorrhage (PPH) (more than 500 ml) and the rate of severe PPH (more than 1000 ml).

The principal outcome of the study is the volume of postpartum blood, this volume is measured by the midwife who is responsible of the birth. Collection of lost blood is initiated immediately after birth of the baby by passing a blood collection drape under the woman's buttocks.

The secondary outcomes are the influence of acupuncture in the placental expulsion time, and the influence of the predictor variables in the bleeding volume and in the placental expulsion time: primiparity or multiparity, number of gestation including abortions, doses of oxytocin during labor, maternal age, maternal weight in the beginning of the gestation, maternal ponderal gain during pregnancy, date of the last blood test during pregnancy and value of hemoglobin and hematocrit, spontaneous labor or induction by means of oxytocin or prostaglandins, spontaneous or artificial rupture of membranes, first stage of labor duration, second stage of labor duration, hours since rupture of membranes, hours since epidural analgesia, volume of serotherapy during labor, and newborn weight. Possible puerperal complications or security problems, the degree of Satisfaction of the Mother and the degree of ease with which the acupuncturist administered the treatment are also secondary outcomes.

DETAILED DESCRIPTION:
This study is designed as a single-blind randomized clinical trial with parallel design, and third party evaluation at the Hospital Universitario Príncipe de Asturias in Alcalá de Henares (Madrid, Spain). The study will be carry out with pregnant women who were in labor at this hospital. Information sheets about the study will be distributed by the different health care centers coordinated by the hospital. The midwives will give the information sheets to pregnant women during the pregnancy's attendances. The objective is to let pregnant women know about the study before their labor date in order to encourage them to participate in it.

Pregnant women fulfilling all the inclusion criteria and none of the exclusion criteria will be invited to participate in the experiment. These requirements includes pregnant women from 18 to 40 years old, with eutectic delivery, gestation between 37 and 42 weeks, labors with epidural analgesia.

Concerning the procedure and data collection, the acupuncturist will request permission to midwife responsible of the mother for their collaboration in the study in the pre-labor room. The acupuncturist will explain the study to the mother and her partner and will apply for her voluntary participation being the informed consent offered then. All information will be given when the pregnant woman is without pain of labor, preferably when the woman is under the epidural analgesia effects.

Regarding to the selection of patients, a randomization scheme will be performed using an envelope based method. The researches will have opaque envelopes with a number outside, this number being the code of the patient in the study. After the approval of the pregnant woman and informed consent, the acupuncturist opens the envelop which will indicate the treatment to follow, either control or intervention group. So, investigators guarantee randomization, blindness and unpredictable selection of the sample.

In the labor ward, after delivery, the baby is placed on the abdomen of the puerperal mother to facilitate maternal link. Collection of lost blood is initiated immediately after birth of the baby by passing a blood collection bag under the woman's buttocks. The birth attendant clamps the umbilical cord at first minute after birth and the acupuncturist midwife performed the acupuncture procedure depending on the group assigned.

In the intervention group with real acupuncture, after the umbilical cord is clamped, the acupuncturist disinfects the abdominal area with antiseptic and pricks the needle in the point Ren Mai 6. In the control group the puncture of the Ren Mai 6 is not performed. In both cases, the needle is covered with a opaque plastic cup and the cup is set with adhesive tape, guaranteeing that both the midwife responsible of the birth and the puerperal woman do not know if the Ren Mai 6 acupuncture point has been punctured or not.

Afterwards, the midwife responsible of the birth expects to note the signs of placental separation such as a gush of blood, uterine contraction, lengthening of the umbilical cord, and visualization of the placenta in the vagina, and then encourage the woman to cough of push. When the placental has been expelled, the midwife pays attention to the time passed from the delivery to the placental expulsion, and she changes the collected bleeding drape for another one if the puerperal women has to be sutured. Finally, a nappy is settled to the puerperal woman until the first two hours after birth. This procedure is routinely used at this hospital.

The midwife responsible of the birth weights one or both blood collection drapes, gauzes used and nappy, and registers the data in a specific record. Taking into account the total weight and the amount of material used, the volume of blood loss is estimated.

A survey will be fulfilled by the acupuncturist no more than 2 hours after the intervention. In this survey, the midwife takes notes on the level of ease with which the technique was performed with four possible answers (high, moderate, medium and low ease level). Furthermore, the acupuncturist will ask to the puerperal woman if she would recommend this technique to any of her friends with two possibles answers (yes or not).

The placental expulsion time will be measured after the childbirth is occurred. The weight of the blood collected drapes, gauzes and nappy is registered in the first two hours after birth, so too, the satisfaction of professionals and participants is noted in this time. After this period of time, the puerperal woman is moved to the obstetrics plant which is out of the labor room. Participants will be followed-up during the hospital stay, an expected average of 2 days. The physician in charge of evaluation of the welfare of the puerperal woman will annotate the existence or not of complications during the hospital stay in the medical record of the woman, as it is routinely done at hospital.

All the study will be performed in conditions of respect for individual rights and ethical principles affecting biomedical research involving human. Written informed consent will be fulfilled by all participants. In particular, the physical and mental integrity of women will be safeguarded, as well as privacy and data protection in accordance to the Spanish Organic Law 15/1999, of December 13, Protection of Personal Data. All the participants will give their informed consent in accordance with the Declaration of Helsinki assuring confidentiality and freedom to withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women from 18 to 40 years old
* Within 37 and 42 gestation weeks
* Low obstetric risk labor
* With epidural analgesia

Exclusion Criteria:

* Pregnant woman with metal allergy
* Patients with anticoagulant treatment
* Dystocic labor
* Uterine overdistension
* Precipitous (less than 2 hours) or prolonged ( more than 11 hours) first stage of labor
* Pregnant woman with coagulation disorders
* Alterations in the placental insertion
* Pregnant woman with curettage
* Woman with previous uterine surgery or myomatosis
* Use of uterine relaxants during labor
* Patients who do not understand Spanish or are not be able to understand the procedure of the study or to sign the informed consent.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Postpartum blood loss | First two hours after birth
  This volume is measured by the midwife responsible of the birth who does not know if the point is punctured or not, thus guaranteeing the third party evaluation.

SECONDARY OUTCOMES:
Placental Expulsion Time | First two hours after birth
  This time is measured by the midwife responsible of the birth, and it is considered as the time passed between the delivery of the newborn and the complete expulsion of the placenta.
Number of participants with puerperal complications | 48 hours after birth
  According to routine procedure, the physician who is in charge of the postpartum unit notes any complications that occurred within 48 hours of the birth on the medical record of the puerperal woman. The items are: Uterine Atony, Placental Retention, Urinary Retention, Postpartum Hemorrhage (>500ml), and Others, with two possible answers (yes or no).
Degree of Satisfaction of the Mother | Two hours after labor
  This item is analyzed by a specific survey that the midwife carries out no more than 2 hours after the labor. The midwife asks to the mother if she would recommend this technique to any of her friends with two possible answer (yes or no).
Degree of ease with which the technique was administered | Two hours after labor
  The acupuncturist completed a survey no more than 2 hours after the intervention. In this survey, the acupuncturist noted the ease with which the acupuncturist administered the treatment (high, moderate, medium, and low ease).

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Lopez Garrido, Midwife, Principal Investigator — Hospital Universitario Principe de Asturias
Locations (1):
- Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid, Spain